CLINICAL TRIAL: NCT00201305
Title: Prospective Phase II Randomized Trial-Weekly Gemcitabine Plus High-Dose 5-Fluorouracil/ Leucovorin in the Treatment of Advanced or Metastatic Carcinoma of the Biliary Tract
Brief Title: Gemcitabine Plus High-Dose 5-Fu/Leucovorin in the Treatment of Advanced or Metastatic Carcinoma of the Biliary Tract
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: Chang Gung Memorial Hospital (Other); Changhua Christian Hospital (Other); China Medical University Hospital (Other); Mackay Memorial Hospital (Other); Chi Mei Medical Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government); National Cheng-Kung University Hospital (Other); National Taiwan University Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T3202
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2009-04-01 (Estimated); Status verified 2005-09

CONDITIONS: Biliary Tract Disease
MeSH Terms: conditions — Biliary Tract Diseases

INTERVENTIONS:
Drug: Gemcitabine+5FU+Leucovorin

SUMMARY:
This is an open-label phase II trial with weekly gemcitabine plus high-dose 5-FU/leucovorin infusion (HDFL) for patients with advanced or metastatic carcinoma of the biliary tract. The primary endpoint is patients' response and the secondary endpoints are chemotherapy-related toxicity, time to disease progression and overall survival. .

DETAILED DESCRIPTION:
5-FU has been the mainstay of chemotherapeutic agents for gastrointestinal malignancies. The use of weekly 24-hour infusion of HDFL produces high clinical response in a variety of cancers, including colorectal, gastric and breast cancers, with minimal chemotherapy-related toxicity. Gemcitabine is a synthesized deoxycytidine analogue that is metabolized to dFdCTP in tumor cells and results in inhibition of DNA synthesis and depletion of normal cellular nucleotide pool. It has been shown to be active in the treatment of pancreatic cancer and non-small cell lung cancer. Since the biliary tract and the pancreas share a common embryonic origin and cancers from both sites are characterized by resistance to most chemotherapeutic agents, we postulate that gemcitabine may also be effective for cancer of the biliary tract. In our institution we have devised a regimen of weekly gemcitabine and 24-hour infusion of HDFL for patients with advanced or metastatic pancreatic adenocarcinoma. In 18 evaluable patients, 2 achieved a partial response and 3 minor response. The median duration of response was 4 months and the treatment-related toxicity was acceptable.

The eligibility criteria are patients with advanced or metastatic carcinoma of the biliary tract who are not candidates for curative surgical treatment; good performance status; no prior chemotherapy; clinical measurable tumor; good organ function and good compliance. Each cycle of chemotherapy consists of 4 weeks. On days 1, 8 and 15, gemcitabine will be given by 30-minute intravenous infusion and 5-FU and leucovorin by 24-hour continuous intravenous infusion. The dose of gemcitabine will be 1000 mg/m2. The doses of 5-FU will be 2000 mg/m2 and leucovorin, 300 mg/m2. Treatment will continue until disease progresses or prohibitive toxicity develops. For patients with complete response (CR), chemotherapy will continue for 3 additional courses after the documentation of CR. Estimated time for patient accrual is 3 years.

ELIGIBILITY:
Inclusion criteria:

1. Histologically proven carcinoma of the biliary tract, including gallbladder carcinoma and cholangiocarcinoma. The disease should be either locally advanced to the extent that curative surgery is impossible or with documented distant metastasis.
2. Bi-dimensionally measurable disease by physical examination or image study (roentgenogram or computed tomography (CT) scan).
3. Age > 18 years. For patients older than 70 years of age, detailed evaluation of the organ function reserves must be done before enrollment unto protocol treatment.
4. Karnofsky performance status> 60%
5. Adequate bone marrow reserves, defined as white blood cell (WBC)>4,000/ml, absolute neutrophil count (ANC)> 1,500/ml, platelet> 150,000/ml.
6. Liver transaminases <5 times upper normal limits; total bilirubin <3 mg/dl; serum creatinine < 1.5 mg/dl
7. Serum triglyceride level >70 mg/dl
8. No prior cytotoxic chemotherapy. Previous radiotherapy is allowed if the treatment was completed at least 6 weeks before the enrollment onto this study.
9. Patients of childbearing age should have effective contraception during the study period.
10. All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional guidelines.

Exclusion criteria:

1. Patients who are receiving concurrent radiotherapy, chemotherapy or other experimental therapy.
2. Patients who refuse port-A catheter implantation
3. Patients with brain or leptomeningeal metastases.
4. Patients who have significant cardiac arrhythmia or acute myocardial infarction within 6 months before entry.
5. Patients who have major systemic diseases that the attending physicians considered inappropriate for systemic chemotherapy.
6. Life expectancy less than 2 months.
7. Pregnant or nursing women may not participate. Women or men with reproductive potential may not participate unless they have agreed to use an effective contraceptive method.
8. Patients who have previous malignancy except for the following: adequately treated basal cell or squamous cell skin cancers, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any cancer from which the patient has been disease-free for 5 years.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2002-07; Study Completion 2012-08

PRIMARY OUTCOMES:
To determine the response rate of weekly gemcitabine plus high-dose 5-FU/leucovorin chemotherapy for patients with advanced or metastatic biliary tract cancer.

SECONDARY OUTCOMES:
To determine:
1.Toxicity profile of gemcitabine plus high-dose 5-FU/leucovorin chemotherapy for advanced or metastatic biliary tract cancer.
2.Time to disease progression
3.Overall survival
4.Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Li Cheng, PHD, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- See also: Related Info — http://english.nhri.org.tw/inst_cancer/ca_TCOGresearch.php